CLINICAL TRIAL: NCT01974843
Title: The Assessment of Bupivacaine-tramadol and Levobupivacaine-tramadol Combinations for Preemptive Caudal Anaesthesia in Children: a Randomized, Double-blind, Prospective Study
Brief Title: Caudal Block With Tramadol and Levobupivacaine or Bupivacaine
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, gulbin sezen, assistant of professor, Duzce University
Other Study IDs: DZC-160
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine; Bupivacaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group BT: Bupivacaine-tramadol (BT) group received a caudal injection of bupivacaine 0.25% plus tramadol 2 mg/kg
  Interventions: Drug: Bupivacaine
- Group LT: Levobupivacaine-tramadol (LT) group received a caudal injection of levobupivacaine 0.25% plus tramadol 2 mg/kg, resulting in a total volume of 1 ml/kg.
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — in the levobupivacaine-tramadol (LT) group received a caudal injection of levobupivacaine 0.25% plus tramadol 2 mg/kg (maximum doses; 35 mg levobupivacaine plus 35 mg tramadol), resulting in a total volume of 1 ml/kg at maximum volume of 15 ml
  Other Names: Chirocaine, Abbott Lab, Nycomed Pharma, Norway
  Groups: Group LT
Drug: Bupivacaine — in the bupivacaine-tramadol (BT) group received a caudal injection of bupivacaine 0.25% plus tramadol 2 mg/kg (maximum doses; 35 mg bupivacaine plus 35 mg tramadol)
  Other Names: Marcaine, Astra Zeneca, UK
  Groups: Group BT

SUMMARY:
Caudal block is the regional anesthetic technique that is used most frequently in pediatric surgery. Opioid drugs have been added to local anesthetic solutions to prolong duration of analgesia but ideal combination were not found that has minimal adverse effect. The aim of this study was to compare the postoperative analgesic efficacy of equal concentrations of bupivacaine plus tramadol or levobupivacaine plus tramadol in pediatric patients undergoing minor urological surgery.

DETAILED DESCRIPTION:
Sixty-eight children aged 2 to 7 years who were undergoing inguinal herniorrhaphy or orchidopexy received bupivacaine 0.25% plus tramadol 2 mg/kg (BT group) or levobupivacaine 0.25% plus tramadol 2 mg/kg (LT group) by the caudal route after laryngeal mask anesthesia. The primary outcome of the study was to compare the duration and quality of postoperative analgesia. The postoperative pain relief was evaluated by the Children and Infants Postoperative Pain Scale (CHIPPS) at 2, 4, 6, 12, and 24 h postoperatively. In addition, the time of first analgesic requirement was noted.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,
* 2 to 7 years old children
* Elective inguinal herniorrhaphy or orchidopexy operation

Exclusion Criteria:

* Infection at the site of block, bleeding diathesis, pre-existing neurological or spinal disease, or abnormalities of the sacrum) or with a known allergy to local anesthetics were excluded.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ASA status I children aged 2 to 7 years who were scheduled for elective inguinal herniorrhaphy or orchidopexy were enrolled.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Quality of postoperative analgesia | Postopertively 24 h
  The postoperative pain relief was evaluated by the Children and Infants Postoperative Pain Scale (CHIPPS) at 2, 4, 6, 12, and 24 h postoperatively. In addition, the time of first analgesic requirement was noted.

SECONDARY OUTCOMES:
Adverse effect | Postoperatively at 2, 4, 6, 12, and 24 h
  All patients were observed in the hospital for at least 24 h because of the possible side effects of caudal blocks.

OTHER OUTCOMES:
first analgesic requirement | Postoperatively 24 h
  In the case of a CHIPPS score of 4 or more, paracetamol 30 mg.kg -1 was administered rectally. The duration of analgesia was defined by noting the time from caudal injection to the time of first analgesic requirement.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University Medicine School, Anesthesiology and Reanimation Department, Düzce, Turkey (Türkiye)

REFERENCES:
- [Background] Silvani P, Camporesi A, Agostino MR, Salvo I. Caudal anesthesia in pediatrics: an update. Minerva Anestesiol. 2006 Jun;72(6):453-9. PMID 16682915
- [Background] Locatelli B, Ingelmo P, Sonzogni V, Zanella A, Gatti V, Spotti A, Di Marco S, Fumagalli R. Randomized, double-blind, phase III, controlled trial comparing levobupivacaine 0.25%, ropivacaine 0.25% and bupivacaine 0.25% by the caudal route in children. Br J Anaesth. 2005 Mar;94(3):366-71. doi: 10.1093/bja/aei059. Epub 2004 Dec 17. PMID 15608043
- [Background] Yildiz TS, Ozdamar D, Bagus F, Solak M, Toker K. Levobupivacaine-tramadol combination for caudal block in children: a randomized, double-blinded, prospective study. Paediatr Anaesth. 2010 Jun;20(6):524-9. doi: 10.1111/j.1460-9592.2010.03296.x. Epub 2010 Apr 14. PMID 20412459
- See also: caudal block usage in pediatric patients — http://www.paccjournal.com/
- See also: performing of caudal block in pediatric patients — http://www.nysora.com/